CLINICAL TRIAL: NCT00001030
Title: A Prospective, Randomized, Comparative Study of the Safety and Efficacy of Clarithromycin Versus Rifabutin Versus the Combination of Clarithromycin Plus Rifabutin for the Prevention of Mycobacterium Avium Complex (MAC) Bacteremia or Disseminated MAC Disease in HIV-Infected Patients With CD4 Lymphocyte Counts <= 100 Cells/mm3
Brief Title: The Safety and Effectiveness of Clarithromycin and Rifabutin Used Alone or in Combination to Prevent Mycobacterium Avium Complex (MAC) or Disseminated MAC Disease in HIV-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 196; CPCRA 009; 11172 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Mycobacterium Avium-intracellulare Infection; HIV Infections
Keywords: Rifabutin; Mycobacterium avium-intracellulare Infection; Acquired Immunodeficiency Syndrome; Clarithromycin
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Clarithromycin; Rifabutin

INTERVENTIONS:
Drug: Clarithromycin
Drug: Rifabutin

SUMMARY:
To compare the efficacy and safety of clarithromycin alone versus rifabutin alone versus the two drugs in combination for the prevention or delay of Mycobacterium avium Complex (MAC) bacteremia or disseminated MAC disease. To compare other parameters such as survival, toxicity, and quality of life among the three treatment arms. To obtain information on the incidence and clinical grade of targeted gynecologic conditions.

Persons with advanced stages of HIV are considered to be at particular risk for developing disseminated MAC disease. The development of an effective regimen for the prevention of disseminated MAC disease may be of substantial benefit in altering the morbidity and possibly the mortality associated with this disease and its treatment.

DETAILED DESCRIPTION:
Persons with advanced stages of HIV are considered to be at particular risk for developing disseminated MAC disease. The development of an effective regimen for the prevention of disseminated MAC disease may be of substantial benefit in altering the morbidity and possibly the mortality associated with this disease and its treatment.

Patients are randomized to receive clarithromycin alone, rifabutin alone, or the two drugs in combination daily. Patients are evaluated every 4 weeks for the first 8 weeks and every 8 weeks thereafter for the duration of the study. Patients are followed for 24 months. Per amendment, a pharmacokinetic substudy will be conducted.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Recommended:

* PCP prophylaxis.

Allowed:

* GM-CSF or G-CSF.
* Erythropoietin.
* Therapies (including antiretrovirals) available through expanded access or treatment IND programs.
* Other non-experimental therapies available by prescription.
* Antihistamines other than those specifically excluded.

Patients must have:

* Evidence or diagnosis of HIV infection or a history of an AIDS-defining condition by CDC criteria.
* CD4 count <= 100 cells/mm3 within 90 days prior to study entry.
* Two baseline blood sample cultures negative for MAC within 30 days of study entry.
* No suspected disseminated MAC disease, in the opinion of the clinician.

NOTE:

* Patients with elevated GGT and/or triglycerides are allowed.

NOTE:

* Patients may co-enroll on ACTG 081/981/181, ACTG 175, ACTG 204, ACTG 193, ACTG 241, or other acceptable protocols.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Known or suspected tuberculous infection or other non-tuberculous mycobacterial infection requiring chemotherapy or chemoprophylaxis (with the exception of isoniazid prophylaxis alone).

NOTE:

* Patients may enroll who successfully completed tuberculosis (TB) treatment and have been off anti-TB drugs for more than 6 months with no symptoms of mycobacterial infection.
* Active TB.
* Known hypersensitivity to study drugs.
* Malabsorption as defined by persistent diarrhea with more than 8 stools per day for > 6 weeks.

Concurrent Medication:

Excluded:

* Frequent (more than once per month), repeated, or continuous treatment courses of quinolones, erythromycin, spiramycin, azithromycin, clarithromycin, or clindamycin.
* Concomitant terfenadine or astemizole.

Prior Medication:

Excluded:

* Prophylaxis with azithromycin, clarithromycin, or rifabutin for more than 4 months.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1100
Dates: Study Completion 1996-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benson CA, Study Chair; Cohn DL, Study Chair
Locations (42):
- United States (41):
  - Alabama Therapeutics CRS, Birmingham, Alabama
  - UCLA CARE Center CRS, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - Ucsf Aids Crs, San Francisco, California
  - Howard University Hosp., Div. of Infectious Diseases, ACTU, Washington D.C., District of Columbia
  - Univ. of Miami AIDS CRS, Miami, Florida
  - Univ. of Hawaii at Manoa, Leahi Hosp., Honolulu, Hawaii
  - Chicago Children's CRS, Chicago, Illinois
  - Northwestern University CRS, Chicago, Illinois
  - Cook County Hosp. CORE Ctr., Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - Methodist Hosp. of Indiana, Indianapolis, Indiana
  - Univ. of Iowa Healthcare, Div. of Infectious Diseases, Iowa City, Iowa
  - Johns Hopkins Adult AIDS CRS, Baltimore, Maryland
  - Massachusetts General Hospital ACTG CRS, Boston, Massachusetts
  - Bmc Actg Crs, Boston, Massachusetts
  - Beth Israel Deaconess - East Campus A0102 CRS, Boston, Massachusetts
  - Beth Israel Deaconess Med. Ctr., ACTG CRS, Boston, Massachusetts
  - Hennepin County Med. Ctr., Div. of Infectious Diseases, Minneapolis, Minnesota
  - University of Minnesota, ACTU, Minneapolis, Minnesota
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - Univ. of Nebraska Med. Ctr., Durham Outpatient Ctr., Omaha, Nebraska
  - SUNY - Buffalo, Erie County Medical Ctr., Buffalo, New York
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Memorial Sloan-Kettering Cancer Ctr., New York, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - Cornell University A2201, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Bronx-Lebanon Hosp. IMPAACT CRS, The Bronx, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Carolinas HealthCare System, Carolinas Med. Ctr., Charlotte, North Carolina
  - Regional Center for Infectious Disease, Wendover Medical Center CRS, Greensboro, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington
- Mbeya Med. Research Program, Mbeya Referral Hosp. CRS, Mbeya, Tanzania

REFERENCES:
- [Background] Currier JS, Williams P, Feinberg J, Becker S, Owens S, Benson CA. ACTG 815: a prospective study of bacterial infections in advanced HIV disease. Conf Retroviruses Opportunistic Infect. 1997 Jan 22-26;4th:131 (abstract no 364)
- [Background] Mascolini M. FDA advisory committee deadlocks on delavirdine. Food and Drug Administration. AIDS Treat News. 1996 Dec 6;(No 260):3-5. PMID 11364022
- [Background] Watts DH, Spino C, Benson C, Yu B, Katzenstein D, Hammer S, Stratton P, Korvick J. A comparison of gynecologic findings in HIV-positive women with CD4 lymphocyte counts 200 to 500/cc and less than 100/cc. Int Conf AIDS. 1996 Jul 7-12;11(2):275 (abstract no ThB4137)
- [Background] Fichtenbaum CJ, Zackin R, Feinberg J, Benson C, Griffiths JK; AIDS Clinical Trials Group New Works Concept Sheet Team 064. Rifabutin but not clarithromycin prevents cryptosporidiosis in persons with advanced HIV infection. AIDS. 2000 Dec 22;14(18):2889-93. doi: 10.1097/00002030-200012220-00010. PMID 11153670
- [Background] Cohn DL. Prevention strategies for Mycobacterium avium-intracellulare complex (MAC) infection. A review of recent studies in patients with AIDS. Drugs. 1997;54 Suppl 2:8-15; discussion 28-9. doi: 10.2165/00003495-199700542-00004. PMID 9358195
- [Background] Watts DH, Spino C, Zaborski L, Katzenstein D, Hammer S, Benson C. Comparison of gynecologic history and laboratory results in HIV-positive women with CD4+ lymphocyte counts between 200 and 500 cells/microl and below 100 cells/microl. J Acquir Immune Defic Syndr Hum Retrovirol. 1999 Apr 15;20(5):455-62. doi: 10.1097/00042560-199904150-00007. PMID 10225227
- [Background] Fichtenbaum CJ, Powderly WG. Refractory mucosal candidiasis in patients with human immunodeficiency virus infection. Clin Infect Dis. 1998 Mar;26(3):556-65. doi: 10.1086/514571. PMID 9524822
- [Background] Benson CA, Williams PL, Cohn DL, Becker S, Hojczyk P, Nevin T, Korvick JA, Heifets L, Child CC, Lederman MM, Reichman RC, Powderly WG, Notario GF, Wynne BA, Hafner R. Clarithromycin or rifabutin alone or in combination for primary prophylaxis of Mycobacterium avium complex disease in patients with AIDS: A randomized, double-blind, placebo-controlled trial. The AIDS Clinical Trials Group 196/Terry Beirn Community Programs for Clinical Research on AIDS 009 Protocol Team. J Infect Dis. 2000 Apr;181(4):1289-97. doi: 10.1086/315380. Epub 2000 Apr 13. PMID 10762562
- [Background] Currier JS, Williams P, Feinberg J, Becker S, Owens S, Fichtenbaum C, Benson C; Adult Clinical Trial Group. Impact of prophylaxis for Mycobacterium avium complex on bacterial infections in patients with advanced human immunodeficiency virus disease. Clin Infect Dis. 2001 Jun 1;32(11):1615-22. doi: 10.1086/320515. Epub 2001 Apr 30. PMID 11340534